CLINICAL TRIAL: NCT01126567
Title: A Study of the Effects of Sampling Rate on Cerebrospinal Fluid (CSF) Biomarker Levels in Healthy Subjects
Brief Title: Exploratory Biomarker Study of Cerebrospinal Fluid in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Daniel LLano, M.D., PhD, Associate Medical Director, Abbott
Other Study IDs: F09-113
Record Dates: First submitted 2010-02-24; First posted 2010-05-19 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
Keywords: Phase 1 Clinical Trials, Cerebrospinal Fluid, Biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, cerebrospinal fluid

GROUPS / COHORTS (2):
- High Sampling Rate: Samples will be obtained at a high rate
  Interventions: Other: Sampling Rate
- Low Sampling Rate: Samples will be obtained at a low rate
  Interventions: Other: Sampling Rate

INTERVENTIONS:
Other: Sampling Rate — Both cohorts will have a lumbar catheter placed and CSF samples will be obtained. The only difference between the two arms will be the sampling rate of CSF. One arm will have a high sampling rate and the other will have a low sampling rate.

SUMMARY:
The objective of this study is to determine the effects of cerebrospinal fluid sampling rate on biomarker levels of young, healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age is between 18 and 50 years, inclusive
* Judged to be in general good health based on medical history, physical exam, neuro exam, vital signs, lab profile and ECG

Exclusion Criteria:

* Positive urine drug screen for drugs of abuse
* History of bleeding disorder or deep vein thrombosis
* History of migraine or other types of headache more than twice/month, history of spinal disc disease or chronic significant low back pain
* Use of blood thinning compounds within 10 days of lumbar drain placement
* Finding on head CT that contraindicates lumbar puncture
* History of spinal surgery
* Use of tobacco/nicotine containing products within 6 month period prior to initial lumbar drain placement

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Multiple Exploratory Biomarkers | Day 1 (at 0, 1, 4, 8, 12, 18, and 24 hours)
Multiple Exploratory Biomarkers | Day 1 (at 0, 1.2.3.4.5.6.7.8.9.10,12,14,16,18,20,22,and 24 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lenz, M.D., Ph.D., Study Director — Abbott
Locations (1):
- Glendale, California, United States